CLINICAL TRIAL: NCT01698450
Title: MR-Guided Functional Ultrasound-Neurosurgery for Movement Disorders
Brief Title: Magnetic Resonance (MR) Guided Functional Ultrasound-Neurosurgery for Movement Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK: 2012-0027
Record Dates: First submitted 2012-07-02; First posted 2012-10-03 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Essential Tremor; Dystonia; Parkinson's Disease
Keywords: FUS; focused ultrasound; functional brain disorder; neuropathic pain; movement disorders; malignant brain tumors
MeSH Terms: conditions — Essential Tremor; Dystonia; Parkinson Disease; Neuralgia; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Focused Ultrasound for Movement Disorders (Other)
  Interventions: Device: Non-invasive intervention with focused ultrasound (ExAblate 4000)

INTERVENTIONS:
Device: Non-invasive intervention with focused ultrasound (ExAblate 4000) — Non-invasive brain intervention using MR-guided focused ultrasound
  Other Names: ExAblate 4000

SUMMARY:
The aim of this study is to asses the efficacy and the clinical safety of the transcranial magnetic resonance guided high intensity focused ultrasound system ExAblate 4000, InSightec Ltd. for functional neurosurgery in the treatment of movement disorders. The treatments to be conducted in this study are non-invasive, i.e. without opening the skull, and will create microthalamotomies in specific target areas such as thalamus, subthalamus and pallidum. The data obtained in this study will be used to evaluate the basic safety aspects of this new treatment technology and will serve as a basis for the clinical introduction of MR-guided ultrasound neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 18 and 80 years, inclusive.
* Patients who are able and willing to give consent and able to attend all study visits.
* A diagnosis of a MD, such as Essential Tremor (ET), Idiopathic Parkinson's diseases or primary Dystonia as confirmed from clinical history and examination by a movement disorder neurologist.
* A MD refractory to adequate medical treatment, or in whom the indication for Deep Brain Stimulation (DBS) would be given, but DBS cannot be performed because of medical comorbidities or medical reasons, or because the patient clearly confirms by written statement that he does not want to undergo DBS for personal reasons (PD: increasing motor fluctuations albeit optimal medical treatment & unbearable side effects of medication; ET: failure of adequate tremor control with Propranolol and Primidone alone and in combination; Dystonia: dystonia or pain not controlled by oral medication). An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
* Either the medial thalamic nuclei or the subthalamic or pallidal areas can be target by the ExAblate device. The target region must be apparent on MRI such that targeting can be performed with either direct visualization or by measurement from landmarks, using the "Stereotactic Atlas of the Human Thalamus and Basal Ganglia" by Anne Morel, 39 analogous to our first clinical FUS study on patients with chronic pain 33.
* Able to communicate sensations during the ExAblate MRgFUS treatment
* Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
* Significant disability due to MD despite medical treatment (speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities)
* Inclusion and exclusion criteria have been agreed upon by two members of the medical team.

Exclusion Criteria:

* Patients with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Patients with documented myocardial infarction within six months of protocol entry
  * Congestive heart failure requiring medication (other than diuretic)
  * Patients on anti-arrhythmic drugs
* Patients exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:

  * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
  * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
  * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
  * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
* Severe hypertension (diastolic BP > 100 on medication)
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium) including advanced kidney disease
* Severely impaired renal function (estimated glomerular filtration rate < 45ml/min/ 1.73 m2) or receiving dialysis
* History of abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Active or suspected acute or chronic uncontrolled infection
* History of intracranial hemorrhage
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
* Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Participation in another clinical trial in the last 30 days
* Patients unable to communicate with the investigator and staff.
* Presence of any other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
* Compromised Immune System, including HIV positive serum status
* Known life-threatening systemic disease
* Patients with a history of seizures within the past year
* Patients with current or a prior history of any psychiatric illness will be excluded. Any presence or history of psychosis will be excluded. Patients with a significant mood disorders including depression will be excluded. For the purpose of this study, we consider a significant mood disorder to include any patient who has:

  * been under the care of a psychiatrist for over 3 months
  * taken antidepressant medications for greater than 6 months
  * has participated in cognitive-behavioral therapy
  * been hospitalized for the treatment of a psychiatric illness
  * received transcranial magnetic stimulation
  * received electroconvulsive therapy
* Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy
* Patients with brain tumors
* Any illness that in the investigator's opinion preclude participation in this study.
* Pregnancy or lactation.
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Lesion Size | 3 months
  Size of lesion in the target area for each sonication as a function of applied energy/temperature.
Patient Safety | 3 months
  Number of Patients with Adverse Events as a Measure of Safety and Tolerability.

SECONDARY OUTCOMES:
Clinical efficacy and QOL | 3 months
  Efficacy and QOL will be quantified on respective rating scales (specified in protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Ernst - Martin, MD, Principal Investigator — University Children's Hospital, Zurich; Ronald - Bauer, MD, Principal Investigator — Neurosurgey, Kantonsspital St. Gallen, Switzerland
Locations (1):
- MR-Center, University Children's Hospital, Zurich, Canton of Zurich, Switzerland